CLINICAL TRIAL: NCT06901479
Title: The Study of Postoperative Delirium and Glymphatic System Function in Cardiac Surgery
Acronym: Delirium
Status: Active, not recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20250225-07
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Delirium (POD)
Keywords: analysis along the perivascular space, diffusion tensor imaging, glymphatic system, Postoperative delirium, cardiac surgery
MeSH Terms: conditions — Emergence Delirium | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Blood samples for proteomic analyses
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- The cardiac surgery postoperative delirium group: 1. Patients who met the inclusion and exclusion criteria underwent MRI assessment of the glymphatic system function before cardiac surgery after signing the informed consent form.
  2. The patients underwent routine cardiac surgery.
  3. Blood was drawn before the surgery.
  4. Delirium was assessed on postoperative days 1 to 5.
  5. Blood was drawn on the second day after surgery, and MRI assessment of the glymphatic system function was performed again on the fifth day after surgery.
  Interventions: Other: Blood was drawn for proteomics testing and Magnetic Resonance Imaging.
- The cardiac surgery postoperative non-delirium group: 1. Patients who met the inclusion and exclusion criteria underwent MRI assessment of the glymphatic system function before cardiac surgery after signing the informed consent form.
  2. The patients underwent routine cardiac surgery.
  3. Blood was drawn before the surgery.
  4. Delirium was assessed on postoperative days 1 to 5.
  5. Blood was drawn on the second day after surgery.
  6. Patients who did not develop postoperative delirium were selected as the control group, matched for age, BMI, and duration of surgery, and underwent MRI assessment of the glymphatic system function again on the fifth day after surgery.
  Interventions: Other: Blood was drawn for proteomics testing and Magnetic Resonance Imaging.

INTERVENTIONS:
Other: Blood was drawn for proteomics testing and Magnetic Resonance Imaging. — The function of the glymphatic system was assessed by MRI before the surgery. Blood was drawn before the surgery. Delirium was assessed on postoperative days 1 to 5. Blood was drawn on the second day after surgery. The function of the glymphatic system was assessed again by MRI on the fifth day after surgery.

SUMMARY:
Postoperative delirium after cardiac surgery is an acute cerebral dysfunction characterized by inattention, impaired consciousness, and cognitive and orientation disturbances. It manifests clinically as acute onset, severe neurocognitive impairment, and periodic fluctuating progression, and is one of the most common complications after major cardiac and vascular surgery. It typically occurs within one week after surgery, with a peak incidence at 24 hours postoperatively. Due to differences in the basic characteristics of study populations and assessment tools, the reported incidence of postoperative delirium after cardiac surgery varies significantly, ranging from 14% to 50%. Postoperative delirium not only prolongs patients' ICU and hospital stays, increases medical costs, and raises short-term and long-term mortality rates, but is also closely associated with long-term cognitive impairment, dementia, and a decline in activities of daily living. The pathophysiology of delirium is complex and may be caused by a combination of multiple factors, including microembolism, ischemia-reperfusion injury, and systemic inflammatory response. Since the mechanisms underlying delirium are not yet fully understood, effective treatments are currently lacking. Postoperative delirium after cardiac surgery is a significant clinical challenge for medical teams.

The brain is distinct from other organs, as the tight junctions of the blood-brain barrier isolate the exchange between the brain, cerebrospinal fluid, blood, and extracellular fluid. For a long time, it was believed that the brain lacks a lymphatic system, and the extracellular fluid in brain tissue was considered stagnant. The lack of fluid flow can lead to the accumulation of protein waste, which is very detrimental to brain health. The glymphatic system is a major update in the anatomical knowledge of the central nervous system in recent years. It is a highly organized fluid transport system within the human brain, with the primary function of promoting convective exchange between the interstitial fluid of the central nervous system and cerebrospinal fluid. The main physiological function of the glymphatic system is to clear metabolic waste and large-molecule solutes, thereby maintaining central homeostasis; it also acts as a communicator between the brain and peripheral immunity, ensuring that the central nervous system is not overlooked by the immune system. Additionally, the glymphatic system helps deliver nutrients to the brain, such as glucose, lactate, and amino acids. Dysfunction of the glymphatic system is associated with various neurological diseases, such as Alzheimer's disease and Parkinson's disease, and related research has become a frontier and hotspot in the field of neuroscience.

Dysfunction of the glymphatic system leads to the accumulation of β-amyloid and tau proteins in the brain, which cannot be cleared, and is one of the pathogenic mechanisms of Alzheimer's disease. There is a strong bidirectional association between Alzheimer's disease and delirium. Patients with Alzheimer's disease-related dementia are 2.5 to 4.7 times more likely to experience delirium, and the incidence of newly diagnosed Alzheimer's disease-related dementia in patients with delirium increases by 12.5 times. However, the underlying mechanisms of postoperative delirium remain unclear, which has motivated our investigation into the causal relationship between the glymphatic system and postoperative delirium. From a theoretical perspective, chronic dysfunction of the glymphatic system signifies brain vulnerability and a higher incidence of neurological diseases. If subjected to surgical stress, sudden dysfunction may represent acute glymphatic system insufficiency. With the rapid development of clinical imaging tools, functional MRI is a non-invasive method for assessing glymphatic system function, bringing possibilities to clinical research.

Therefore, this study aims to explore the association between postoperative delirium after cardiac surgery and the glymphatic system, in order to deepen the understanding of glymphatic system function and investigate the mechanisms of postoperative delirium after cardiac surgery, and to provide ideas for new interventions for postoperative delirium after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing elective cardiac surgery with cardiopulmonary bypass (such as coronary artery bypass grafting, bioprosthetic valve replacement, valve repair, congenital heart surgery, etc.);
2. Age ≥ 60 years.

Exclusion Criteria:

1. Aortic dissection and other surgeries involving major blood vessels;
2. A history of mental illness with related medication use; preoperative Mini-Mental State Examination (MMSE) score < 27; preoperative delirium;
3. A history of neurosurgery or traumatic brain injury; if a focal brain lesion larger than 3 cm occurs during the study, the data will be excluded from subsequent analyses;
4. Hearing and language impairments that affect communication;
5. Contraindications to MRI (e.g., presence of metal implants in the body, including prosthetic valve replacement, internal fixation plates after fracture surgery, etc.).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age over 60 years, undergoing cardiac surgery.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium | Postoperative delirium was assessed on postoperative days 1 to 5
  Using the 3-Minute Diagnostic Assessment for Delirium

SECONDARY OUTCOMES:
Analysis along the perivascular space (ALPS) | 1、Before surgery；2、On the fifth day after surgery
  MRI indicators for assessing glymphatic system function
Blood was drawn for proteomics testing | 1、Before surgery; 2、On the fifth day after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No